CLINICAL TRIAL: NCT02205554
Title: A Phase 1 Randomized, Double-Blind, Placebo-Controlled, Triple Cross-Over Study Investigating The Safety, Oral Steady-State Pharmacokinetics, And Clinical Activity Of 20 Mg Omnitram And 50 Mg Tramadol In Normal Human Subjects
Brief Title: Omnitram Pharmacokinetic Study In Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Syntrix Biosystems, Inc. (Industry)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: Syntrix-Omni-Pain-101; R44DA027304 (NIH)
Record Dates: First submitted 2014-07-28; First posted 2014-07-31 (Estimated); Last update posted 2014-10-15 (Estimated); Status verified 2014-10

CONDITIONS: Pain
Keywords: Analgesia; Pharmacokinetics; Treatment
MeSH Terms: conditions — Pain; Agnosia | interventions — Tramadol

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Omnitram-Tramadol-Placebo (Active Comparator): Omnitram 20 mg every 6 hours for 9 doses, followed by Tramadol 50 mg every 6 hours for 9 doses, followed by Placebo every 6 hours for 9 doses.
  Interventions: Drug: Omnitram; Drug: Tramadol; Drug: Placebo
- Tramadol-Placebo-Omnitram (Active Comparator): Tramadol 20 mg every 6 hours for 9 doses, followed by Placebo every 6 hours for 9 doses, followed by Omnitram 20 mg every 6 hours for 9 doses.
  Interventions: Drug: Omnitram; Drug: Tramadol; Drug: Placebo
- Placebo-Omnitram-Tramadol (Active Comparator): Placebo every 6 hours for 9 doses, followed by Omnitram 20 mg every 6 hours for 9 doses, followed by Tramadol 50 mg every 6 hours for 9 doses.
  Interventions: Drug: Omnitram; Drug: Tramadol; Drug: Placebo

INTERVENTIONS:
Drug: Omnitram — Nine 20 mg doses administered every 6 hours
Drug: Tramadol — Nine 50 mg doses administered every 6 hours.
Drug: Placebo — Nine doses administered every 6 hours.

SUMMARY:
The purpose of this study is to compare the safety, pharmacokinetic properties (the absorption, distribution and excretion), and analgesic activity of Omnitram (10 mg tablets), Tramadol (Ultram, 50 mg tablet) following oral administration of 9 doses healthy subjects.

DETAILED DESCRIPTION:
A Phase 1, single-center, randomized, double-blind, placebo-controlled, three-period cross-over study to compare the safety, steady-state oral pharmacokinetics, and clinical activity of overencapsulated: 20 mg Omnitram (2x10 mg tablets), 50 mg Tramadol (1x50 mg Ultram tablet), and placebo.

Forty male subjects in normal health, 21 to 55 years of age, will be randomized to three parallel arms (N=~13 each) to ingest a total of 9 doses of Omnitram, Tramadol, or placebo in a first treatment segment (one dose every 6 hours). Around the 9th dose blood samples are collected to quantify plasma Tramadol and Metabolite 1 (M1) enantiomers. After the 9th dose, pain tolerance is assessed with a cold pressor test (ice cold water immersion). After the 7th dose abuse liability measures and pupil diameter will be assessed. Subjects will washout for 7 days after the first treatment segment and second treatment segment.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy male with normal vital signs: systolic blood pressure > 90 mm Hg and < 140 mm Hg; diastolic blood pressure > 50 mm Hg and < 90 mm Hg; pulse 50 to 100 beats per minute; respiratory rate 12 to 20 breathes per minute
2. Between the ages of 21 and 55 years of age
3. Able and willing to give informed consent
4. Able to comply with all study procedures
5. Have adequate hematologic function as evidenced by the following screening results:

   * White Blood Cell (WBC) >3,500/mm3 and < 12,000/mm3;
   * Platelet Count > 150,000/mm3 and < 540,000/mm3;
   * Hemoglobin > 12.5 gm/dL and < 20.5 gm/dL.

   Have adequate liver function as evidenced by the following screening results:
   * Aspartate transaminase (AST) ≤ 60 IU/L;
   * Alanine transaminase (ALT) ≤ 83 IU;
   * Alkaline Phosphatase ≤ 150 IU/L;
   * Total Bilirubin ≤ 1.2 mg/dL;
   * Prothrombin Time (PT) < 1.2 upper limit of normal (ULN); Partial Thromboplastin Time (PTT) < 1.2 ULN.
6. Electrocardiogram (ECG) within normal limits as determined by the PI
7. Have adequate renal function as evidenced by the following screening result:

   Glomerular filtration rate (GFR) calculated by Cockcroft-Gault formula >60 ml/min.

   Urinalysis demonstrating < +1 glucose, +1 ketones, and +1 protein
8. Negative urine test for substances of abuse, including opiates, per clinical research unit (CRU) standards
9. Negative serology tests for HIV, hepatitis B surface antigen and hepatitis C virus antibody
10. Body Mass Index (BMI) 19.0 to 32 kg/m
11. Cold pressor screening results as follows: 1) pain tolerance of > 20 seconds and <120 seconds

Exclusion Criteria:

1. Oral temperature > 38°C or history of current illness
2. History of seizures, epilepsy, or recognized increase risk of seizure (e.g., head trauma, metabolic disorders, alcohol or drug withdrawal)
3. History of cirrhosis or laboratory evidence of liver disease
4. Use of alcohol within 24 hours of day -1 until the end of the study; and grapefruit, grapefruit-related citrus fruits (e.g., Seville oranges, pomelos), or grapefruit juice or grapefruit-related juices, or other medication, within 7 days of study drug administration and until the end of the study
5. History of previous anaphylaxis, severe allergic reaction to Tramadol, codeine, or other opioid drugs
6. Use of monoamine oxidase (MAO) inhibitors (including linezolid), Serotonin Reuptake Inhibitors, Serotonin-Norepinephrine Reuptake Inhibitors, and prescription or over-the counter (OTC) medications known to induce or inhibit drug metabolism, including cytochrome P450 2D6 (CYP2D6), and other drugs that may affect the serotonergic neurotransmitter systems including, but not limited to, triptans, dextromethorphan, tricyclic antidepressants, bupropion, lithium, tramadol, dietary supplements such as tryptophan and St. John's Wort, and antipsychotics or other dopamine antagonists. These restrictions are to be maintained from 14 days before study day -1, until the subject completes the study
7. Any other unstable acute or chronic disease that could interfere with the evaluation of the safety of the study drug as determined by the principal Investigator in dialogue with the Sponsor Medical Monitor
8. Unlikely to comply with the study protocol
9. Known or suspected alcohol or drug abuse within the past 6 months
10. Received another investigational agent within 4 weeks of Day 0, or within five half-lives of Day 0, whichever is longer; or receiving any other investigational agent during this study
11. Any concurrent disease or condition that in the opinion of the investigator impairs the subject's ability to complete the trial. Psychological, familial, sociological, geographical or medical conditions which, in the Investigator's opinion, could compromise compliance with the objectives and procedures of this protocol, or obscure interpretation of the trial data

Ages: 21 Years to 55 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 43 (Actual)
Dates: Start 2014-08; Primary Completion 2014-10 (Actual); Study Completion 2014-10 (Actual)

PRIMARY OUTCOMES:
Omnitram and Tramadol Steady State Maximum and Minimum Concentrations | 0.0, 1.0, 1.5, 2.0, 2.5, and 4.0 hours after the 9th dose of Omnitram and Tramadol.
Adverse events | 29 days

SECONDARY OUTCOMES:
Cold Water Induced-Pain Reported On a 0 to 10 Scale | On Study Day 2, Study Day 12, and Study Day 22, after the 9th dose of Omnitram, Tramadol, and placebo.
  Subject immerses a hand in cold water for a maximum of 3 minutes and reports level of pain.
Abuse Liability Assessed With Visual Analogue Scales | On Study Day 1, Study Day 11, and Study Day 21, after the 7th dose of Omnitram, Tramadol, and placebo.
  Subjects read a question and respond by placing a mark on a visual analogue scale.

OTHER OUTCOMES:
Pupil Size | On Study Day 1, Study Day 11, and Study Day 21, after the 7th dose of Omnitram, Tramadol, and placebo.
  A pupilometer is used to measure eye pupil size.

CONTACTS AND LOCATIONS:
Overall Officials: Shawn Searle, MD, Principal Investigator — PRA/CRI Lifetree Research Center; Stuart Kahn, MD, Study Director — Syntrix Biosystems, Inc.
Locations (1):
- CRI Lifetree Research Center, Salt Lake City, Utah, United States

REFERENCES:
- [Derived] Zebala JA, Searle SL, Webster LR, Johnson MS, Schuler AD, Maeda DY, Kahn SJ. Desmetramadol Has the Safety and Analgesic Profile of Tramadol Without Its Metabolic Liabilities: Consecutive Randomized, Double-Blind, Placebo- and Active Comparator-Controlled Trials. J Pain. 2019 Oct;20(10):1218-1235. doi: 10.1016/j.jpain.2019.04.005. Epub 2019 Apr 18. PMID 31005596